CLINICAL TRIAL: NCT02885077
Title: Effects of High-intensity Inspiratory Muscle Training Associated With Aerobic and Resistance Exercise in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Effects of High-intensity Inspiratory Muscle Training in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Isabella Martins de Albuquerque, Effects of high-intensity inspiratory muscle training in patients undergoing coronary artery bypass grafting surgery, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16149813.3.0000.5346
Record Dates: First submitted 2016-08-21; First posted 2016-08-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Complications Due to Coronary Artery Bypass Graft

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-intensity IMT + combined exercise (Experimental): Participants will perform 12 weeks of IMT strength training is achieved with a device with linear load pressure with a device with linear load pressure (POWERbreathe Medic Plus ®, SP, BR). Training will progress to 80% maximal inspiratory pressure (PiMax). IMT will perform for 12 weeks with two sessions per week. The training protocol will consists of five series with ten repetitions with two minutes or according to patient feedback using the modified Borg scale.The initial charge of training will be 50% of PiMax in the first 2 weeks, with an increase of 55% of PiMax in the 3 week, 60% of PiMax in the 4 week, 65% of PiMax in the 5 week, 70% of PiMax in the 6 week, 75% of PiMax in the 7 week and 80% of PiMax in the 8 week. After the 9 and 12 week training period, the PiMax measurements will be performed weekly to keep 80% of the new PiMax.
  Interventions: Device: High-intensity IMT + combined exercise
- H-IMT sham + combined exercise (Sham Comparator): Participants will perform 12 weeks of IMT strength training is achieved with a device with linear load pressure with a device with linear load pressure (POWERbreathe Medic Plus ®, SP, BR). The sham group will perform for 12 weeks with two sessions per week. The protocol will consists of five series with ten repetitions with two minutes and will train at a constant inspiratory load of no more than 10% of their initial Pimax.
  Interventions: Device: High-intensity IMT + combined exercise

INTERVENTIONS:
Device: High-intensity IMT + combined exercise
  Other Names: Sham Control H-IMT + combined exercise

SUMMARY:
Even with the advances in clinical therapy and percutaneous interventions, coronary artery bypass grafting (CABG) is still widely used in the treatment of patients with coronary artery disease (CAD). However, it is a complex procedure that triggers important organic implications especially on pulmonary function. In relation to the treatment of patients undergoing CABG, the recovery is linked to the cardiac rehabilitation programs. These programs can also be associated with other muscle training measures, among these there is inspiratory muscle training (IMT). Most studies has been implemented moderate-intensity IMT daily, but there are few studies about the effects of high intensity training loads performed on alternate days. In this context, is justified the use of a device such as the recent Powerbreathe, which uses higher training loads that would provide greatest benefits, whereas the magnitude of the response to training tends to increase with load.

OBJECTIVE: To investigate the efficiency of high intensity IMT associated with combined aerobic and resistance training on maximal exercise capacity, submaximal exercise capacity, respiratory muscle strenght, pulmonary function, oxidative stress, quality of life and endothelial function in patients who underwent CABG in phase II cardiac rehabilitation program.

METHODOLOGY: This is a clinical trials, controlled, randomized,double-blind being developed in partnership with Cardiology Clinic of Hospital Universitário de Santa Maria (HUSM), Santa Maria, RS, Brazil. Patients will undergo the evaluation of pulmonary function and respiratory muscle strength (spirometry and digital manovacuometry), as well on the maximal exercise capacity (Ergospirometry), submaximal functional capacity (6MWT and 6MST), of quality of live (MLHFQ) of Oxidative stress and endothelial function (blood biomarkers). After the evaluation will be randomly allocated into two groups: the control group will perform cardiac rehabilitation associated with the Sham of IMT, and the experimental group cardiac rehabilitation associated with the IMT High-intensity. The intervention will last twelve weeks for both groups and after this phase patients will be submitted again to the assessment tools.

EXPECTED RESULTS: The high intensity IMT potentiates the effects of cardiac rehabilitation (phase II) after coronary artery bypass surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CABG up to three weeks before the initiation of the study, a clinical course without complications during hospitalization
* Clinically stable
* The absence of smoking (previous or current).

Exclusion Criteria:

* Unstable angina
* Myocardial infarction and heart surgery up to three months before the survey;
* Chronic respiratory diseases
* Hemodynamic instability
* Orthopedic and neurological diseases that may preclude the achievement of the cardiopulmonary test and Cardiac Rehabilitation exercises
* Psychological and / or cognitive impairments that restrict them to respond to questionnaires.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Effects of high-intensity inspiratory muscle training on the functional capacity assessed by cardiopulmonary exercise test (CPT) and measured by VO2 peak. | Finalized study (12 weeks)

SECONDARY OUTCOMES:
Effects of high-intensity inspiratory muscle training on the inspiratory muscle endurance evaluated by using the traditional manovacuometry and the PowerBreathe device. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on lung function assessed by spirometry. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the submaximal functional assessed by six-minute walk test (6MWT) and measured with six minute walk distance. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the submaximal functional capacity assessed by six-minute step test (6MST) and measured with the number of steps. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the quality of life assessed by Minnesota Living with Heart Failure questionnaire (MLHFQ) | Finalized study (12 weeks)
  The MLHFQ is a questionnaire validated for the Brazilian population, consisting of 21 questions regarding limitations frequently associated with the extent to which heart failure has affected patient's lives in the previous month. Each question is attributed a value from 0 (zero) to 5 (five), with the highest score indicating worse quality of life. The total score is calculated by adding the 21 items, with a possible interval between 0 and 105.
Effects of high-intensity inspiratory muscle training on the oxidative stress assessed by analysis of advanced oxidation protein products (AOPP). Plasma levels of AOPP assessed by on automated analyzer Mindray® expressed as µmol/L. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the oxidative stress assessed by analysis of products of ferric reducing antioxidant power (FRAP). Plasma levels of FRAP assesssed by automated analyzer Mindray® expressed as µmol/L. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the endothelial function assessed by analysis of nitric oxide (NOx). Plasma levels of NOx assessed automated analyzer Mindray® expressed as µmol/L. | Finalized study (12 weeks)
Effects of high-intensity inspiratory muscle training on the Inflammatory profile assessed by through ultra-sensitive C-reactive protein (us-CRP) on automated analyzer Mindray® expressed as mg/dL | Finalized study (12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dos Santos TD, Pereira SN, Portela LOC, Cardoso DM, Lago PD, Dos Santos Guarda N, Moresco RN, Pereira MB, de Albuquerque IM. Moderate-to-high intensity inspiratory muscle training improves the effects of combined training on exercise capacity in patients after coronary artery bypass graft surgery: A randomized clinical trial. Int J Cardiol. 2019 Mar 15;279:40-46. doi: 10.1016/j.ijcard.2018.12.013. Epub 2018 Dec 10. PMID 30581100